CLINICAL TRIAL: NCT06731049
Title: Comparison of the Effects of Treadmill-Based Walking and Dual-Task Walking Training on Activity and Cognition in Alzheimer's Disease
Brief Title: Comparison of the Effectiveness of Treadmill-Based Walking and Dual-Task Walking Training in Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kübra Nur Menengiç, MSc, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DT Treadmill Training in AD
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer' Disease; Dementia
Keywords: Treadmill; Dual-task; Exercise; Rehabilitation; Physiotherapy and rehabilitation
MeSH Terms: conditions — Disease; Dementia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill Based Training Group (Active Comparator): In the study, for 8 weeks, the Treadmill-based Training Group will undergo walking training on a treadmill two days a week.
  Interventions: Other: Treadmill-based Training Group
- Dual-Task Treadmill Based Training Group (Experimental): Dual-Task Treadmill-based Training Group will receive dual-task walking training involving both motor and cognitive tasks on the treadmill for 8 week, two days in a week.
  Interventions: Other: Dual-Task Treadmill-based Training Group

INTERVENTIONS:
Other: Treadmill-based Training Group — The walking speed will start at 75% of the walking speed calculated from the 10-meter Walk Test at normal walking pace, and the treadmill training will begin at this speed. Every two weeks, the speed will increase by 5%, and by the end of the 8th week, it will reach 100% of the normal walking speed. The aim of gradually increasing the walking speed is to progressively make the motor component of the exercise more challenging. Throughout the 8 weeks, a body weight support system will be used, and the support from the treadmill bar will be gradually reduced.
  Arms: Treadmill Based Training Group
Other: Dual-Task Treadmill-based Training Group — In the Dual-Task Treadmill-based Training Group, the same walking training protocol as the Treadmill Training Group will be applied with added second tasks to create a dual-task walking protocol. The second tasks will consist of both cognitive and motor tasks. The difficulty of the tasks and the total duration of the dual-task training will be increased over time.
  Arms: Dual-Task Treadmill Based Training Group

SUMMARY:
Alzheimer's disease is a neurodegenerative condition that affects both cognitive and motor functions, making daily life activities more challenging. Motor functions, especially walking and balance, begin to deteriorate early in the disease and progress in parallel with cognitive decline. Dual-task performance, which refers to the ability to perform both motor and cognitive tasks simultaneously, significantly decreases in individuals with Alzheimer's disease. Current studies suggest that dual-task exercises can improve both cognitive and motor functions. In this context, treadmill-based dual-task training emerges as a promising approach to mitigate the effects of Alzheimer's disease. The study hypothesizes that treadmill-based dual-task training will have more positive effects on motor and cognitive parameters compared to treadmill exercise alone in individuals with Alzheimer's disease. The main research question of this study is whether treadmill-based dual-task exercise training, designed with progressively more challenging cognitive and motor tasks and tailored to the individual, results in significant improvements in motor and cognitive parameters, as well as daily living activities and dual-task performance, compared to a group that only undergoes treadmill exercise.

DETAILED DESCRIPTION:
The aim of this project is to investigate the effects of treadmill-based dual-task exercise training, which is individually designed and progressively challenging, on functional mobility, cognitive function, walking speed, balance, and dual-task performance in Alzheimer's disease. The results obtained from this training will be compared only to those of treadmill-based walking training. The goal of this project is to enhance the level of independence in daily life by improving cognitive and physical parameters related to body structure and function. In the study, for 8 weeks, the Treadmill-based Training Group will receive walking training on the treadmill twice a week, while the Dual-Task Treadmill-based Training Group will undergo dual-task walking training, which includes both motor and cognitive tasks on the treadmill. At the beginning and end of the 8-week training period, functional mobility, cognitive function, ability to perform activities of daily living, balance, walking speed, and dual-task performance will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Alzheimer's disease according to the NINCDS-ADRDA criteria by a neurologist,
2. In the early or middle stages of the disease according to the Clinical Dementia Rating Scale (CDR),
3. Receiving medical treatment for Alzheimer's disease (e.g., cholinesterase inhibitors or memantine) for at least the past month,
4. Able to walk at least 400 meters in the 6-Minute Walk Test, indicating functional mobility,
5. Able to read and understand instructions given in Turkish.

Exclusion Criteria:

1. Having Lewy body dementia, frontotemporal dementia, or other types of dementia
2. Participating in a structured exercise program within the 6 months prior to starting the study
3. Having pulmonary, neurological, musculoskeletal, or rheumatological diseases that hinder walking
4. Having an unstable medical condition (e.g., uncontrolled diabetes or hypertension, deep vein thrombosis, etc.)
5. Having visual or auditory impairments that make communication difficult
6. Having behavioral problems that make participation in exercise difficult

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test | From enrollment to the end of treatment at 8 weeks
  Timed Up and Go Test (TUG) In the Timed Up and Go Test, the participant is instructed to stand up from a fixed chair placed on a non-slip surface with their knees and hips at approximately 90 degrees, walk 3 meters, turn around, and sit back down. The time taken to complete these activities is recorded.
Trail Making Test | From enrollment to the end of treatment at 8 weeks
  The Trail Making Test, used to assess executive functions, has two versions: A and B. In version A, a page with scattered numbers is given to the participant, and they are asked to connect the numbers from 1 to 25 in sequence as quickly as possible. In version B, a page with both numbers (1-13) and letters (A-L) is provided. The participant is instructed to connect the numbers and letters in sequence, alternating between 1-A-2-B-3-C, and so on. The time taken to complete each task is recorded in seconds.
Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) | From enrollment to the end of treatment at 8 weeks
  The ADCS-ADL, developed specifically for Alzheimer's disease, consists of 23 items-6 basic and 17 instrumental activities of daily living-that assess the participant's level of independence. Questions are directed to the caregiver, focusing on the participant's performance over the last 4 weeks. The total score ranges from 0 to 78, with lower scores indicating higher levels of dependency.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | From enrollment to the end of treatment at 8 weeks
  MoCA is a widely used screening test for global cognitive function. It assesses cognitive abilities in 6 domains: calculation, abstract thinking, orientation, executive function, memory, verbal fluency, attention, and visual-spatial abilities. A total score above 21 indicates normal cognitive function.
Verbal Fluency Test | From enrollment to the end of treatment at 8 weeks
  The Verbal Fluency Test evaluates verbal fluency and executive functions under two categories: phonemic and semantic fluency. In the phonemic fluency section, the number of words starting with the letters K, A, and S produced by the participant is recorded. In the semantic fluency section, the total number of words related to selected categories such as animals, fruits, furniture, or vehicles is recorded. The total time for the test is 60 seconds, and the number of words produced every 15 seconds is recorded separately.
Digit Span Test | From enrollment to the end of treatment at 8 weeks
  This test is used to assess short-term memory and attention. In the forward digit span section, the participant is asked to repeat the numbers read aloud by the examiner in the same order, while in the backward digit span section, they must repeat the numbers in reverse order. The test begins with a span of 3 numbers, and after correctly repeating the given sequence, the length of the number sequence is increased one digit at a time (e.g., 3-7, 1-5-9, 4-8-2-7, 6-3-1-9-2).
Four-Step Balance Test | From enrollment to the end of treatment at 8 weeks
  This test is used to measure static balance. The participant is asked to stand for 10 seconds in four different positions on a firm and stable surface: with both feet together, semi-tandem, tandem, and one foot.
10-Meter Walk Test | From enrollment to the end of treatment at 8 weeks
  The 10-Meter Walk Test is a performance-based test used to evaluate walking speed. A 14-meter distance is measured, with an additional 2 meters at the start and end of the walking path. The time taken to walk the 10-meter distance is recorded in seconds.
Dual-Task Performance | From enrollment to the end of treatment at 8 weeks
  Dual-task performance will be assessed by applying the Timed Up and Go Test along with cognitive tasks such as naming animals, generating words starting with the same letter, and repeating given sequences of numbers in order.

IPD SHARING:
Plan to Share IPD: No